CLINICAL TRIAL: NCT01100398
Title: Prevalence of Nonalcoholic Fatty Liver Disease and Nonalcoholic Steatohepatitis Utilizing Ultrasound and Percutaneous Liver Biopsy: A Prospective Cohort Study
Brief Title: Prevalence of Nonalcoholic Fatty Liver Disease (NAFLD) and Nonalcoholic Steatohepatitis (NASH) Utilizing Ultrasound and Percutaneous Liver Biopsy
Status: Completed | Type: Observational
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Christopher D. Williams, MD (fellow, gastroenterology), Brooke Army Medical Center
Other Study IDs: Williams-NASH1
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Fatty Liver
Keywords: Fatty liver disease
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — liver biopsies and serum blood samples may be obtained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NAFLD/NASH prevalence: Any subject between the ages of 18-70 without known fatty liver disease who meet inclusion criteria
  Interventions: Procedure: possible liver biopsy and serum collection

INTERVENTIONS:
Procedure: possible liver biopsy and serum collection — All patients with a positive ultrasound for hepatic steatosis offered a liver biopsy after obtaining fasting blood work that included a complete blood count, coagulation studies, liver function tests, fasting lipid panel, glucose and insulin. Patients with a negative ultrasound for fatty liver are not referred for liver biopsy and are considered as completed study patients. Serum is also stored for adipokine and cytokine analysis. A study investigator using a 14g Bard Monopty biopsy gun performs the liver biopsy.

SUMMARY:
Prospective determination of the prevalence of non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH)in a primary care setting using ultrasound and percutaneous liver biopsy.

DETAILED DESCRIPTION:
Patients between the ages of 18 and 70 years who are eligible for care at Brooke Army Medical Center are considered for enrollment. After obtaining informed consent, a baseline questionnaire is given to patients who present to the Primary Care Clinic for routine clinic visits or during colon cancer screening classes within the Gastroenterology Clinic. The questionnaire includes information about the patient's past medical history to include: known history of chronic liver disease, current medications, current and past alcohol ingestion, dietary habits that included consumption of fructose containing beverages and frequency of fast food visits. Patients are excluded if they are found to have a history of chronic liver disease, HIV, on medications that are associated with a fatty liver, or consumption of more than 20 grams of alcohol per day. Right upper quadrant ultrasound will then be performed to determine if there is evidence of fatty liver disease. All patients with a positive ultrasound for hepatic steatosis are then offered a liver biopsy after obtaining fasting blood work that included a complete blood count, coagulation studies, liver function tests, fasting lipid panel, glucose and insulin. Patients with a negative ultrasound for fatty liver are not referred for liver biopsy and are considered as completed study patients. Serum is also stored for adipokine and cytokine analysis. A study investigator using a 14g Bard Monopty biopsy gun will perform the liver biopsy. A single expert hepatopathologist will review all liver biopsies and utilize the Brunt system (9) for grading and staging of steatohepatitis if present.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 70 years of age were recruited from the Primary Care Clinics or the Gastroenterology Clinic at Brooke Army Medical Center. After completing a baseline questionnaire, all patients had a right upper quadrant ultrasound. If fatty liver was identified, then laboratory data and a liver biopsy were obtained.

Exclusion Criteria:

* ETOH consumption over 20 grams/day
* known fatty liver disease, chronic liver disease, HIV, or medication ingestion associated with fatty liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 to 70 years of age who have access to care through the Primary Care Clinics or the Gastroenterology Clinic at Brooke Army Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Study Director — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Derived] Williams CD, Stengel J, Asike MI, Torres DM, Shaw J, Contreras M, Landt CL, Harrison SA. Prevalence of nonalcoholic fatty liver disease and nonalcoholic steatohepatitis among a largely middle-aged population utilizing ultrasound and liver biopsy: a prospective study. Gastroenterology. 2011 Jan;140(1):124-31. doi: 10.1053/j.gastro.2010.09.038. Epub 2010 Sep 19. PMID 20858492